CLINICAL TRIAL: NCT01809067
Title: The Effects of Lavender Aromatherapy on the Reduction of Stress and Anxiety During MRI Procedures. A Randomized Study Comparing the Use of Lavender Aromatherapy to no Aromatherapy.
Brief Title: The Effects of Lavender Aromatherapy on Reducing Stress and Anxiety During MRI Procedures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3887-2
Record Dates: First submitted 2013-03-04; First posted 2013-03-12 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2013-03

CONDITIONS: Anxiety
Keywords: stress; anxiety; MRI; aromatherapy
MeSH Terms: conditions — Anxiety Disorders | interventions — lavender oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lavender Aromatherapy Inhalers (Active Comparator): Lavender Aromatherapy Inhalers
  Interventions: Other: Lavender aromatherapy inhalers
- No aromatherapy (No Intervention): No aromatherapy

INTERVENTIONS:
Other: Lavender aromatherapy inhalers — Patients will self-administer lavender aromatherapy from hand held inhalers containing lavender essential oil.
  Other Names: LAVENDER Essential Oil (Lavendula angustifolia)
  Arms: Lavender Aromatherapy Inhalers

SUMMARY:
Research Question:

What effect if any does the use of lavender aromatherapy have on a patient's stress and anxiety during the MRI procedure in the Cardiovascular Services Department?

Hypothesis:

1. The use of lavender aromatherapy will reduce anxiety by 20% during MRI procedures.
2. MRI cancellations related to stress and anxiety will decrease by 10%.

Sample size of 30 patients is needed for the control group and the lavender aromatherapy group, for a total of 60 patients.

Rationale:

Patients undergoing MRI procedures may experience stress and anxiety related to the small and confining space required during the scan. Anyone with a history of claustrophobia, panic attacks, or fear of enclosed spaces is more likely to experience symptoms of panic, fear, or anxiety during the MRI procedure (Harris, Cumming, & Menzies, 2004, p. 1). This stress and anxiety may cause the patient to abort the scan, the patient may refuse future scans, or the patient's nervous tremors or involuntary quivering may adversely affect the images obtained. Lavender aromatherapy has been shown to reduce stress and anxiety for patients in other settings; however, its use during MRI procedures has not been studied.

This project investigates the use of lavender aromatherapy as a non-pharmacological way to help patients relax during their MRI procedure. Lavender aromatherapy has been studied and shown to reduce stress and anxiety for patients in other situations, but it has not been studied during MRI procedures. Lavender is known to be uplifting, as well as soothing and helpful for reducing stress, anxiety, depression, and insomnia (Herz, 2007, p. 264). If aromatherapy proves useful as an agent to reduce stress and anxiety, patient satisfaction with their MRI procedure will increase and the need for sedating medication could decrease.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Able to voluntarily provide consent
* Undergoing elective MRI procedure

Exclusion Criteria:

* Lavender sensitivity or allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Comparison between patients using aromatherapy and those without aromatherapy | Within one hour following the MRI procedure
  A comparison will be made between the two groups, one group using lavender aromatherapy and one group without aromatherapy. T-tests will be used to assess whether the two groups are statistically different from each other.
  Comparisons will be made by using information collected from the patient with this screening tool: (Patients will complete the screening tool before and after their MRI procedure.)
  State Trait Anxiety Scale (State portion only)

SECONDARY OUTCOMES:
The number of MRI cancellations related to patient stress and anxiety will be compared between the aromatherapy group and those without aromatherapy. | Up to 16 weeks
  A simple comparison will be made using the percentage of cancellations in each group of patients, the group using aromatherapy and those without aromatherapy.
Comparison between patients using aromatherapy and those without aromatherapy | Within one hour following the MRI procedure
  A comparison will be made between the two groups, one group using lavender aromatherapy and one group without aromatherapy. T-tests will be used to assess whether the two groups are statistically different from each other.
  Comparisons will be made by using information collected from the patient with this screening tool: (Patients will complete the screening tool before and after their MRI procedure.)
  Perceived Stress Scale
Comparison between patients using aromatherapy and those without aromatherapy | Within one hour following the MRI procedure
  A comparison will be made between the two groups, one group using lavender aromatherapy and one group without aromatherapy. T-tests will be used to assess whether the two groups are statistically different from each other.
  Comparisons will be made by using information collected from the patient with this screening tool: (Patients will complete the screening tool before and after their MRI procedure.)
  Visual Analog Scale for anxiety - VAS, 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Carol H Machemer, BSN, Principal Investigator — Allina Health System
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Harris LM, Cumming SR, Menzies RG. Predicting anxiety in magnetic resonance imaging scans. Int J Behav Med. 2004;11(1):1-7. doi: 10.1207/s15327558ijbm1101_1. PMID 15194514
- [Background] Herz RS. Aromatherapy facts and fictions: a scientific analysis of olfactory effects on mood, physiology and behavior. Int J Neurosci. 2009;119(2):263-90. doi: 10.1080/00207450802333953. PMID 19125379